CLINICAL TRIAL: NCT03165266
Title: Incremental Role of 2 Dimensional Speckle Tracking Echocardiography in Diagnosis of Right Ventricular Involvement in Patients With Inferior Wall Myocardial Infarction Undergoing Primary Percutaneous Coronary Intervention
Brief Title: Right Ventricular Involvement in Inferior Myocardial Infarction Patients Using 2 Dimensional Speckle Tracking Echocardiography
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, EGAbdelrhman, principal investgator, Assiut University
Other Study IDs: RVINFMI
Record Dates: First submitted 2017-05-19; First posted 2017-05-24 (Actual); Last update posted 2017-05-24 (Actual); Status verified 2017-05

CONDITIONS: Acute Myocardial Infarction of Inferior Wall Involving Right Ventricle (Disorder)
MeSH Terms: interventions — Echocardiography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Two dimensional Echocardiography — I- Routine transthoracic assessment for Left Atrium and Left Ventricle dimensions :
  II- transthoracic assessment of the Right ventricular systolic function by:
  1. . Right Ventricle fractional area change.
  2. . Tricuspid annular plane systolic excursion .
  3. . Tissue Doppler derived tricuspid annular systolic velocity.
  4. . Right ventricle myocardial performance index . III- Assessment of Right ventricular diastolic function: is carried out by pulsed Doppler of the tricuspid inflow, or tissue Doppler of the lateral tricuspid annulus.
  IV Assessment of Right Ventricle chamber quantification:
  * Right ventricular basal, mid ,and longitudinal dimensions.
  * Right ventricular Outflow Tract, and wall thickness V- Assessment of right atrial major ,and minor dimensions ,and right atrial End- systolic area IV- Assessment of longitudinal Right ventricular strain and strain rate by speckle tracking

SUMMARY:
Right ventricular infarction usually occurs in association with inferior myocardial infarction in about 10-50% of the cases. Currently the presence of elevation in right pericordial leads is the most powerful indicator of right ventricular infarction.

The incidence of right ventricular infarction is more in postmortem studies,meaning that Right ventricular infarction is underestimated, possible explanation for this difference could be explained that electrocardiographic sign of Right ventricular infarction disappear early or patients presented late.

DETAILED DESCRIPTION:
The incidence of right ventricular infarction is more in postmortem studies,meaning that Right ventricular infarction is underestimated, possible explanation for this difference could be explained that electrocardiographic sign of Right ventricular infarction disappear early or patients presented late

The role of Right ventricular systolic function in inferior myocardial infarction patients with or without Right ventricular infarction Had been studied. In our study we will Assess Right Ventricular infarction in patients of acute inferior myocardial infarction undergoing primary percutaneous coronary intervention by correlating electrocardiogram, Right ventricular systolic function by echocardiography with the angiographic finding.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of recent acute inferior myocardial infarction.
2. Patients managed by Primary percutaneous coronary intervention.

Exclusion Criteria:

1. Pervious inferior Myocardial Infarction.
2. Inferior Myocardial Infarction treated by thrombolytic therapy.
3. Chronic pulmonary disease.
4. estimatedPulmonary Artery Systolic Pressure ≥35 mmHg by Echocardiography.
5. Valvular heart disease. 6- Dilated cardio-myopathy patients.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: the study include patients with Acute inferior Myocardial in Assuit University Hospital in the duration beginning from June 2017 .
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-06-01 (Estimated); Primary Completion 2018-01-01 (Estimated); Study Completion 2018-02-28 (Estimated)

PRIMARY OUTCOMES:
Right ventricular dysfunction | 3days
  right ventricular dysfunction by Echocardiography as indicator of right ventricular infarction in inferior wll myocardial patients

CONTACTS AND LOCATIONS:
Overall Officials: Marwa M Abdelmohsen, Lecturer, Study Chair — Assiut University

REFERENCES:
- [Background] Andersen HR, Nielsen D, Falk E. Right ventricular infarction: larger enzyme release with posterior than with anterior involvement. Int J Cardiol. 1989 Mar;22(3):347-55. doi: 10.1016/0167-5273(89)90276-3. PMID 2707915
- [Background] Andersen HR, Falk E, Nielsen D. Right ventricular infarction: frequency, size and topography in coronary heart disease: a prospective study comprising 107 consecutive autopsies from a coronary care unit. J Am Coll Cardiol. 1987 Dec;10(6):1223-32. doi: 10.1016/s0735-1097(87)80122-5. PMID 3680789
- [Background] Wagner GS, Macfarlane P, Wellens H, Josephson M, Gorgels A, Mirvis DM, Pahlm O, Surawicz B, Kligfield P, Childers R, Gettes LS, Bailey JJ, Deal BJ, Gorgels A, Hancock EW, Kors JA, Mason JW, Okin P, Rautaharju PM, van Herpen G; American Heart Association Electrocardiography and Arrhythmias Committee, Council on Clinical Cardiology; American College of Cardiology Foundation; Heart Rhythm Society. AHA/ACCF/HRS recommendations for the standardization and interpretation of the electrocardiogram: part VI: acute ischemia/infarction: a scientific statement from the American Heart Association Electrocardiography and Arrhythmias Committee, Council on Clinical Cardiology; the American College of Cardiology Foundation; and the Heart Rhythm Society. Endorsed by the International Society for Computerized Electrocardiology. J Am Coll Cardiol. 2009 Mar 17;53(11):1003-11. doi: 10.1016/j.jacc.2008.12.016. No abstract available. PMID 19281933
- [Background] Javed S, Rajani AR, Govindaswamy P, Radaideh GA, Abubaraka HA, Qureshi TI, Arshad HB. Right ventricular involvement in patients with inferior myocardial infarction, correlation of electrocardiographic findings with echocardiography data. J Pak Med Assoc. 2017 Mar;67(3):442-445. PMID 28303997
- [Background] Zornoff LA, Skali H, Pfeffer MA, St John Sutton M, Rouleau JL, Lamas GA, Plappert T, Rouleau JR, Moye LA, Lewis SJ, Braunwald E, Solomon SD; SAVE Investigators. Right ventricular dysfunction and risk of heart failure and mortality after myocardial infarction. J Am Coll Cardiol. 2002 May 1;39(9):1450-5. doi: 10.1016/s0735-1097(02)01804-1. PMID 11985906
- [Background] O'Rourke RA, Dell'Italia LJ. Diagnosis and management of right ventricular myocardial infarction. Curr Probl Cardiol. 2004 Jan;29(1):6-47. doi: 10.1016/j.cpcardiol.2003.08.003. No abstract available. PMID 14872197
- [Background] Bayata S, Avci E, Yesil M, Arikan E, Postaci N, Tuluce SY. Tricuspid annular motion in right coronary artery-related acute inferior myocardial infarction with or without right ventricular involvement. Anadolu Kardiyol Derg. 2011 Sep;11(6):504-8. doi: 10.5152/akd.2011.134. Epub 2011 Jul 25. PMID 21788200
- [Background] Rudski LG, Lai WW, Afilalo J, Hua L, Handschumacher MD, Chandrasekaran K, Solomon SD, Louie EK, Schiller NB. Guidelines for the echocardiographic assessment of the right heart in adults: a report from the American Society of Echocardiography endorsed by the European Association of Echocardiography, a registered branch of the European Society of Cardiology, and the Canadian Society of Echocardiography. J Am Soc Echocardiogr. 2010 Jul;23(7):685-713; quiz 786-8. doi: 10.1016/j.echo.2010.05.010. No abstract available. PMID 20620859